CLINICAL TRIAL: NCT06326476
Title: An Open-label Parallel Group Pilot Study to Demonstrate the Safety and Efficacy of Subcutaneous Siplizumab in the Treatment of Hidradenitis Suppurativa
Brief Title: An Open-label, Time-lagged, Dose-escalation Study to Evalaute the Safety and Efficacy of Subcutaneous Siplizumab in the Treatment of Hidradenitis Suppurativa.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: ITB-Med LLC (Industry)
Responsible Party: Principal Investigator, Tiffany Mayo, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012699; 000544067 (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — siplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- siplizumab 10mg (Experimental): Up to 6 participants may receive a 10 mg subcutaneous dose of siplizumab from week 0 to week 4 then at weeks 6 and 8.
  Interventions: Drug: Siplizumab
- siplizumab 20mg (Experimental): Up to 6 participants may receive a 20 mg subcutaneous dose of siplizumab from week 0 to week 4 then at weeks 6 and 8.
  Interventions: Drug: Siplizumab
- siplizumab 40mg (Experimental): Up to 6 participants may receive a 40 mg subcutaneous dose of siplizumab from week 0 to week 4 then at weeks 6 and 8.
  Interventions: Drug: Siplizumab

INTERVENTIONS:
Drug: Siplizumab — 40 mg doses

SUMMARY:
This study is to investigate the efficacy of siplizumab in the treatment of Hidradenitis Suppurativa.

DETAILED DESCRIPTION:
Subjects will be assigned to receive seven subcutaneous doses of siplizumab over an 8 week period. The study will include up to 3 investigational treatment cohorts, 10 mg, 20 mg and a 40 mg cohort. Each cohort will contain from 3-6 subjects. The cohort will be administered either 10 mg, 20mg, or 40mg siplizumab SC weekly from baseline (week 0) to week 4 and a dose at weeks 6 and 8. Assessments will be performed weekly from baseline (week 0) through week 6 and biweekly through week 12 (weeks 8, 10 & 12) by an investigator. Weeks 5 and 10 will be telephone visits and will not include physician HS assessments. All other visits will be conducted in person. During all visits, subjects will also be asked to complete a quality of life questionnaire (DLQI) and Visual Analog Scale (VAS) for pain assessment.

A total enrollment of 12 subjects is anticipated in this pilot study; however, up to 18 patients may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age, and provide informed consent prior to study procedures.
* Have moderate to severe HS classified as Hurley stage II or III for at least 6 months refractory to conventional therapies with a total AN count of greater than or equal to 5 prior to enrollment/randomization
* Failed at least 1 course of oral antibiotics for treatment of HS (or demonstrated intolerance to, or had a contraindication to oral antibiotics for treatment of their HS).
* Women of Childbearing potential must have a urine pregnancy test at screening, wk 0 and prior to administration of the study medication
* Women of childbearing potential must be willing to continue a highly effective method of birth control throughout the study (oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal foam/gel/film/cream/suppository (if available in their locale); male partner sterilization (the vasectomized partner should be the sole partner for that participant); true abstinence (when this is in line with the preferred and usual lifestyle of the participant).
* Negative screening for tuberculosis (TB) (Quantiferon Gold, T-spot) within 3 months prior to screening
* If a positive history of latent tuberculosis:

  * Currently receiving treatment for latent TB per standard of care
  * Have documentation of having completed treatment within 5 years prior to baseline
* Agree not to have a live vaccination during the study.

Exclusion Criteria:

* Any other active skin disease that in the opinion of the investigator would interfere with the assessment of HS
* Have greater than 20 draining fistulas at screening or Day 1 prior to enrollment/randomization
* Receipt of non-biologic treatments for HS within 4 weeks prior to baseline other than antibiotics or hormonal therapy
* Receipt of biologic agents within 3 months prior to baseline
* Receipt of any other investigational product within 3 months prior to baseline
* Receipt of new oral antibiotics or hormonal therapy within 6 weeks prior to baseline.

  * Subjects may be included if they are on steady dose of doxycycline or tetracycline antibiotics only for at least 6 weeks prior to baseline visit and may not change or discontinue dose during course of study.
* Receipt of intralesional kenalog injections within 2 weeks prior to baseline
* Any uncontrolled diagnosis or condition that in the opinion of the investigator will interfere with the assessments or the study.
* Currently has a malignancy or a history of a malignancy within 5 years before screen (except successfully treated non-melanoma skin cancer or cervical carcinoma in situ)
* History of an ongoing, chronic or recurrent infectious disease
* Are currently pregnant, breastfeeding, or planning to get pregnant during the study.
* Previous hypersensitivity reaction to siplizumab or to any of the components
* Known infection with HIV, hepatitis B or hepatitis C at screening or randomization.

Patients who are Hepatitis B Core antibody and/or Hep B Surface Antigen positive will be excluded from this study. Patients who are Hepatitis C ab positive will also be excluded from this study.

* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy.
* Any of the following laboratory abnormalities within 30 days of enrollment:

  * White blood count (WBC) < 3 x 103/μL;,
  * CD4+ count below the lower limit of normal,
  * Platelet count < 150,000 /μL,
  * Hemoglobin < 10 g/dL,
  * ALT ≥ 2x upper limit of normal (ULN) or
  * AST ≥ 2x ULN
  * Serum creatinine >1.5x ULN in adults.
  * Positive molecular testing of SARS-CoV-2
  * ALC less than 800 lymphocytes/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | Weeks 4, 8 and 12
  Inflammatory lesions are defined as inflammatory nodules or abscesses. These will be counted at screening, baseline, weeks 1-4, then at week 6 and 8. We will then asses the average change in inflammatory lesion count per subjects at weeks 4, 8 and 12.

SECONDARY OUTCOMES:
Change in Hidradenitis Suppurativa Clinical Response (HiSCR) | Weeks 4,8, and 12.
  The HiSCR assessment is utilized to show clinical improvement. It is a set of 3 criteria where relative to baseline, each has to be met in order to consider a person's Hidradenitis Suppurativa to be improving. This criteria are as follows:
  1. >50% reduction in the total number of inflammatory nodules and abscesses
  2. No increase in abscess count
  3. No increase in draining fistula count
Change in Hurley Stage | Weeks 4,8, and 12
  The Hurley Staging system characterizes the extent of disease in patients with HS. The stages are as follows with 1 having the least involvement and 3 having the most involvement.
  Stage I: Single of multiple abscess formation without sinus tracts and cicatrization Stage II: Recurrent single or multiple abscesses, widely separated, with limited sinus tracts and cicatrization Stage III: Diffuse or near-diffuse involvement of multiple interconnected tracts and abscesses across an entire area
Change in Dermatology Life Quality Index (DLQI) scores | Weeks 4, 8, and 12
  The DLQI is a validated general dermatology questionnaire that consists of 10 items that assess subject health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). Each item has a choice of 4 responses ('not at all', 'a little', 'a lot', and 'very much'. The corresponding scores are '0', '1', '2', or '3'. The total score is the sum of the score of each question. The higher the total score the more a patient's life is affected by their skin condition.
Improvement in Visual Analogue Scale (VAS) pain scores | Weeks 4, 8, and 12
  A 10-point visual analog pain scale will be used with 0 equaling 'no pain' and 10 equaling 'the worst possible pain'.
Change in Lesion Counts | Weeks 4, 8, and 12
  All lesions will be counted and examined at each visit to see if there has been a change in the number of lesions from the previous study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Mayo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States